CLINICAL TRIAL: NCT06268561
Title: Ozurdex Endophtamitis Cohort, Prognostic Assessment at 12 Months
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN852023/CHUSTE
Record Dates: First submitted 2023-11-16; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Endophthalmitis
Keywords: OZURDEX; Visual Acuity; Endophtalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OZURDEX patients: Patients treated by Dr Garcin and Pr Thuret CHU of Saint Etienne in the context of post-OZURDEX endophthalmitis
  Interventions: Other: Visual acuity analysis; Other: Intraocular pressure analysis; Other: Analysis of optical coherence tomography (OCT) images; Other: Analysis of retinograms

INTERVENTIONS:
Other: Visual acuity analysis — Collection of information on visual acuity from the medical file concerning the surgery
Other: Intraocular pressure analysis — Collection of information on intraocular pressure from the medical file concerning the surgery
Other: Analysis of optical coherence tomography (OCT) images — Collection and analysis of optical coherence tomography (OCT) images of the medical file concerning the surgery
Other: Analysis of retinograms — Collection and analysis of retinography images of the medical file concerning the surgery

SUMMARY:
OZURDEX endophthalmitis is a rare and potentially very serious pathology. Different treatments can be carried out early and change the functional prognosis of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had endophtalmitis following an OZURDEX implant injection within 2 months

Exclusion Criteria:

* Intra oculaire procedure in the interval between the injection of OZURDEX and endophtalmitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by Dr Garcin and Pr Thuret CHU of Saint Etienne in the context of post-OZURDEX endophthalmitis
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 2018 to 2023
  Evolution of visual acuity from the first to the last patient includes

SECONDARY OUTCOMES:
IOP measured in mmHg by tonometer and confirmed with Goldman Applanation | 2018 to 2023
  Changes intra ocular pressure.
Tomography | 2018 to 2023
  Changes in the outer retina on optical coherence tomography
Resumption of intravitreal therapy | 2018 to 2023
  Number of new intravitreal injections necessary to control the princeps pathology (AMD/OMD...) during the follow-up of the study ; i.e. relapse of activity of the princeps pathology

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud GARCIN, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No